CLINICAL TRIAL: NCT06990022
Title: Carbohydrate Mouth Rinse Reduces Perceived Exertion and Mental Fatigue, and Improves Technical Actions During Small-Sided Soccer Games
Brief Title: Carbohydrate Mouth Rinse (Small-Sided Soccer Games)
Acronym: CHOMR-SSGs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ersan Arslan, Prof. Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UGaziosmanpasa-2
Record Dates: First submitted 2025-05-12; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Performance; Soccer; Carbohydrate; Mental Fatigue; Technical Skill
Keywords: Game-based training; Carbohydrate; Game performance; Psychophysiological; Performance analysis
MeSH Terms: conditions — Mental Fatigue | interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were strictly separated and think their intervention is the main intervention. The same was true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHO Mouth Rinse Protocol (CHO-MR) (Experimental): CHO solution was a maltodextrin-based mixture containing 6.4% maltodextrin (Protein Ocean, Türkiye). An CHOMR was performed prior to SSGs.
  Interventions: Other: Carbohydrate
- Placebo Protocol (Experimental): The PLA solution consisted of pure water. A mouth rinse was performed before the SSGs.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Carbohydrate — CHO solution was a maltodextrin-based mixture containing 6.4% maltodextrin (Protein Ocean, Türkiye). An CHOMR was performed prior to SSGs. The solution was sweetened with non-caloric artificial sweeteners consisting of sucralose. The CHO solution was prepared in an equivalent saccharin base and shaken for 30 seconds in a vortex mixer to ensure distinguishability. Participants swished the solution in their mouth for 10 seconds before SSGs and then emptied it back into the container to be weighed again. To ensure that the solutions were not swallowed, the containers were measured before and after all MRs using a full precision balance (Etekcity, USA) accurate to 1 g/0.04 oz
  Arms: CHO Mouth Rinse Protocol (CHO-MR)
Other: Placebo — The PLA solution consisted of purified water. Both solutions were made indistinguishable by adding 50 mg of non-calorific artificial sweetener and 50 mg of sucralose (Fibrelle, Turkey). A 25 ml bolus of 6.4% maltodextrin solution was used in a pre-weighed plastic container and sucralose water was tested as PLA for each rinse solution.
  Arms: Placebo Protocol

SUMMARY:
The present study evaluated the influence of carbohydrate mouth-rinsing (CHO- MR) and placebo (PLA) conditions on the psychophysiological responses, kinematic profiles, and technical performance of young male soccer players in 4-Small sided games (SSGs). The study participants were involved in a randomized, double-blind, repeated-measures design that employed 3 sessions (familiarization, CHOMR and PLA) over fifteen days at a testing facility. Participants took part in two test sessions one week apart. CHO solution was a maltodextrin-based mixture containing 6.4% maltodextrin (Protein Ocean, Türkiye). The PLA solution consisted of pure water. Both solutions were made indistinguishable by incorporating 50 mg of a non-calorific artificial sweetener and 50 mg og sucralose (Fibrelle, Türkiye). A 25-ml bolus of 6.4% maltodextrin solution was utilized in a pre-weighed plastic cup, with sucralose water tested as PLA for each rinse solution.

DETAILED DESCRIPTION:
The current study used a double-blind, randomized, and counterbalanced crossover design to compare the effects of CHOMR or PLA on psychophysiological, kinematic responses and technical actions during 4-a-side SSGs. The study intervention programs lasted the same time of the day during separate training sessions in the in-season to avoid various chronobiological factors. The average temperature was 30 °C, with a relative humidity of 35% of the baseline assessments. Second assessments were recorded that the average temperature was 31 °C with a 35% relative humidity. Before the SSGs sessions, anthropometric characteristics were assessed. Players also completed the Yo-Yo Intermittent Recovery Test level 1 (YYIRTL-1) to balance the groups and equally distribute players among SSGs teams based on maximal oxygen uptake ( 2max). The order of different SSGs (CHOMR or PLA) and solutions (MR or PLA) was determined by randomization (www.randomization.com). Each SSGs was separated at least one week apart to minimize the potential negative impact of physical and psychological fatigue on game performance. Continuous monitoring and recording of the heart rate (HR), rating of perceived exertion (RPE), enjoyment and mental fatigue (MF), kinematic responses, and technical actions were conducted during all SSGs. Mood responses were assessed before and after each SSGs. UEFA A licenced strength and conditioning coaches consistently implemented all SSGs sessions on an artificial soccer pitch with verbal coach encouragement.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male soccer players
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Being under 14 years old
* Having a chronic disease
* Contraindication for carbohydrate mouth-rinsing (CHO-MR)

Ages: 14 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
Psychophysiological Responses-Heart Rate | From baseline to the end of treatment at 2 weeks
  Participants used a Polar H10 heart rate (HR) transmitter synchronized with a Polar V800 watch to track the HR throughout the session. Participants' heart rate mean, heart rate peak and heart rate percentage were recorded.
Psychophysiological Responses-Rating of Perceived Exertion | From baseline to the end of treatment at 2 weeks
  Exercise intensity in all test sessions was quantified using the rating of perceived exertion (RPE), which employs a category ratio scale ranging from 6 to 20. This scale has recently been applied in sports psychology to assess effort related to emotions and performance during competitive events.
Psychophysiological Responses-Enjoyment-Brunel mood of states | From baseline to the end of treatment at 2 weeks
  All participants completed the Exercise Enjoyment Scale (EES), which consists of eight items rated on a 1-7 Likert scale. This scale has been validated to measure the enjoyment of exercise in Turkish adolescents and adults. 1 indicates no enjoyment and 7 indicates enjoyment.
Psychophysiological Reactions-Mood Rating | From baseline to the end of treatment at 2 weeks
  A scale consisting of 24 items and six (6) subscales (anger, confusion, depression, fatigue, tension and vitality) was used in all testing sessions. The depression subscale of the scale is an indicator of depressed mood rather than clinical depression. C in all test sessions. The depression subscale of the scale is an indicator of depressed mood rather than clinical depression Participants were asked the question 'How are you feeling right now?' before and after the games and were asked to tick a number between 0 and 4 (0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, 4 = extremely).
Psychophysiological Responses-Mental Fatigue Assessment | From baseline to the end of treatment at 2 weeks
  All test sessions were assessed using the MF visual analogue scale (VAS). The VAS is a subjective rating scale that assesses an individual's perception or experience of a particular construct, such as fatigue. To measure MF using the VAS, individuals are typically presented with a horizontal line or scale with one end zero (0) meaning "no fatigue" or "not tired at all" and the other end one hundred (100) meaning "extremely tired" or "very tired". Participants are then asked to place a mark on the line indicating their perceived level of MF.
Evaluating the total distance (TD) | From baseline to the end of treatment at 2 weeks
  During the SSG sessions, total distance (TD)data were recorded using a Global Navigation Satellite System (GNSS) with a frequency of 10 Hertz and a triaxial accelerometer (STATSports, Apex, Northern Ireland) with a frequency of 100 Hertz. All data recorded by the GNSS units were downloaded and processed using STAT Sports Software (Apex version 3.0.02011).
Assessment of high intensity running distance (HIMD) | From baseline to the end of treatment at 2 weeks
  During the SSG sessions, high-intensity running distance (HIMD) data were recorded using a Global Navigation Satellite System (GNSS) with a frequency of 10 Hertz and a triaxial accelerometer (STATSports, Apex, Northern Ireland) with a frequency of 100 Hertz. All data recorded by the GNSS units were downloaded and processed using STAT Sports Software (Apex version 3.0.02011).
Evaluation of sprint (SD) | From baseline to the end of treatment at 2 weeks
  During the SSG sessions, sprint (SD) data were recorded using a Global Navigation Satellite System (GNSS) with a frequency of 10 Hertz and a triaxial accelerometer (STATSports, Apex, Northern Ireland) with a frequency of 100 Hertz. All data recorded by the GNSS units were downloaded and processed using STAT Sport Software (Apex version 3.0.02011).
Evaluating acceleration (ACC) and deceleration (DCC) | From baseline to the end of treatment at 2 weeks
  During the SSG sessions, acceleration (ACC) and deceleration (DCC) data were recorded using a Global Navigation Satellite System (GNSS) with a frequency of 10 Hertz and a triaxial accelerometer (STATSports, Apex, Northern Ireland) with a frequency of 100 Hertz. All data recorded by the GNSS units were downloaded and processed using STAT Sport Software (Apex version 3.0.02011).

SECONDARY OUTCOMES:
Anthropometric Measurements 1 | Baseline
  Before breakfast, participants had their weight (kg) measured using a body composition analyser (BC-418MA, Tanita Corp., Tokyo, Japan). This device utilises bioelectrical impedance technology using multiple frequencies (ranging from 1 kHz to 50 kHz) to comprehensively assess body composition parameters.
Anthropometric Measurements 2 | Baseline
  Before breakfast, participants had their height (cm) measured using a body composition analyser (BC-418MA, Tanita Corp., Tokyo, Japan). This device utilises bioelectrical impedance technology using multiple frequencies (ranging from 1 kHz to 50 kHz) to comprehensively assess body composition parameters.
Anthropometric Measurements 3 | Baseline
  Before breakfast, participants had their body mass index (kg/m2) measured using a body composition analyser (BC-418MA, Tanita Corp., Tokyo, Japan). This device utilises bioelectrical impedance technology using multiple frequencies (ranging from 1 kHz to 50 kHz) to comprehensively assess body composition parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Erdinc Gorgulu, Doctorate, Principal Investigator — Tokat Gaziosmanpasa University; Yusuf Soylu, Doctorate, Study Chair — Tokat Gaziosmanpasa University; Ersan Arslan, Doctorate, Study Chair — Tokat Gaziosmanpasa University; Bulent Kilit, Doctorate, Study Chair — Tokat Gaziosmanpasa University; Neil D. Clarke, Doctorate, Study Chair — Birmingham City University; Haitham Jahrami, Doctorate, Study Chair — Ministry of Health, Manama, Bahrain; Achraf Ammar, Doctorate, Study Chair — Johannes Gutenberg University Mainz
Locations (1):
- Tokat Gaiosmanpasa University, Tokat Province, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soylu Y, Chmura P, Arslan E, Kilit B. The Effects of Carbohydrate Mouth Rinse on Psychophysiological Responses and Kinematic Profiles in Intermittent and Continuous Small-Sided Games in Adolescent Soccer Players: A Randomized, Double-Blinded, Placebo-Controlled, and Crossover Trial. Nutrients. 2024 Nov 15;16(22):3910. doi: 10.3390/nu16223910. PMID 39599695
- [Background] Soylu Y, Ramazanoglu F, Arslan E, Clemente FM. Effects of mental fatigue on the psychophysiological responses, kinematic profiles, and technical performance in different small-sided soccer games. Biol Sport. 2022 Oct;39(4):965-972. doi: 10.5114/biolsport.2022.110746. Epub 2021 Dec 30. PMID 36247954